CLINICAL TRIAL: NCT00990405
Title: Phase 4 Study of Helicobacter Pylori Eradication Therapy
Brief Title: Clinical Study to Evaluate the Efficacy and the Safety of Eradication Therapy for Helicobacter Pylori in Functional Dyspepsia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Korean College of Helicobacter and Upper Gastrointestinal Research (Other)
Responsible Party: Seol, Sang-Young/President, Korean Society of Helicobacter and Upper Gastrointestinal Research
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KoreanCHUGR05
Record Dates: First submitted 2009-10-05; First posted 2009-10-06 (Estimated); Last update posted 2009-10-06 (Estimated); Status verified 2009-10

CONDITIONS: Functional Dyspepsia; Helicobacter Pylori Infection
Keywords: Rome III criteria

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lansoprazole+Clarithromycin+Amoxycillin (Experimental): Lansoprazole 30 mg bid, for 7 days Clarithromycin 500 mg bid, for 7 days Amoxicillin 1000 mg bid, for 7 days
  Interventions: Drug: Lansoprzole+Amoxicillin+Clarithromycin

INTERVENTIONS:
Drug: Lansoprzole+Amoxicillin+Clarithromycin — Lansoprazole 30 mg bid, for 7 days Clarithromycin 500 mg bid, for 7 days Amoxicillin 1000 mg bid, for 7 days

SUMMARY:
The role of Helicobacter pylori infection in functional dyspepsia remains controversial. Several randomized controlled trials in western countries have shown no significant advantage over placebo. But some recent studies in Asian population were different compared to the result of studies in the Western population. At the present time, it seems to be difficult to conclude the efficacy of the H.pylori eradication therapy in patients with H. pylori-infected functional dyspepsia.

The investigators hypothesize that eradication of Helicobacter pylori has a sustained global symptom improvement in patients with H. pylori infected functional dyspepsia.

DETAILED DESCRIPTION:
Functional dyspepsia: diagnosed by Rome III criteria of Functional gastrointestinal disorder Treatment regimen: Combination of proton pump inhibitor, Amoxicillin, Clarithromycin for 7 days Placebo: Same shaped placebo drugs

ELIGIBILITY:
Inclusion Criteria:

* Functional dyspepsia by Rome III criteria
* Normal endoscopic findings
* H. pylori positive by Urea breath test

Exclusion Criteria:

* Patients with severe concomitant systemic disease
* Patients with GI surgery
* Females with pregnancy or breast-feeding
* Irritable bowel syndrome, inflammatory bowel disease
* Duodenal Ulcer, Gastric Ulcer, GI bleeding
* History of eradication therapy of Helicobacter pylori
* Malignancy
* Psychosomatic disease

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2009-10; Primary Completion 2010-09 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Global symptom improvement after eradication of Helicobacter pylori in patients with functional dyspepsia therapy) | Symptom assessment at 8 weeks after eradication

SECONDARY OUTCOMES:
To improves the quality of life | 1 year
Global symptom improvement, at 4 weeks after Helicobacter pylori eradication therapy | 1 year
The improvement of 8 dyspeptic symptom | 1 year
The adequate relief of symptom | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Sang-Young Seol, Professor, Study Chair — Korean Society of Helicobacter and Upper Gastrointestinal Research
Locations (1):
- Korean Society of Helicobacter and Upper GI Research, Seoul, Seoul, South Korea